CLINICAL TRIAL: NCT00706901
Title: Impact of Group Motivational Interviewing for Dually Diagnosed Veterans
Brief Title: Impact of Group Motivational Interviewing and In-Home-Messaging-Devices for Dually Diagnosed Veterans
Acronym: GMI-IHMDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDA-2-016-08S; IIR 13-317-2 (Other Grant/Funding Number: Clinical Science Research and Development)
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Alcohol Dependence; Dual Diagnosis; Drug Dependence
Keywords: MI; IHMD
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 GMI (Experimental): Patients randomized to GMI received four structured 75-minute sessions consistent with the central principles and style of motivational interviewing (Miller & Rollnick, 2012). The goal of MI is to develop a sense of discrepancy between personal goals and current behavior and enhance change talk among participants, particularly for taking responsibility of one's substance use and being proactive for remaining in treatment.
  Interventions: Behavioral: Arm 1 GMI; Behavioral: Arm 3 TCC
- Arm 2 IHMD (Experimental): Participants randomized to In-Home-Messaging Devices (IHMD) received a 27-day Care Coordination Home Telehealth (CCHT) program targeting their acute recovery from alcohol and other substance use disorder. Participants received their IHMD device through the Charleston VAMC CCHT program, including device accessories and a phone number to reach their CCHT provider. They were provided with specific instructions on how to set up their IHMD in their residence after discharge. The research associate followed-up with the patient one day after receiving the device to ensure that the device was successfully set up and to provide assistance as necessary. Participants received standard VA CCHT services.
  Interventions: Behavioral: Arm 2 IHMD; Behavioral: Arm 3 TCC
- Arm 3 TCC (Active Comparator): Participants randomized to the Treatment Control Condition (TCC) received a psycho-educational group (e.g., addiction as a chronic disease, relapse prevention, developing a plan to prevent relapse) that was delivered with the aid of sequential standardized PowerPoint presentations. Group members were encouraged to ask questions and make comments. Therapists were encouraged to conduct the sessions using an instructional quality that minimized the use of GMI strategies. TCC consisted of four sessions, lasting 75 minutes, and was conducted on four consecutive days within the course of one week.
  Interventions: Behavioral: Arm 3 TCC

INTERVENTIONS:
Behavioral: Arm 1 GMI — Participants randomized to GMI received four structured, back-to-back, 75-minute sessions in one week consistent with the central principles and spirit of MI (Miller & Rollnick 2013) and based on a manualized protocol (Martino & Santa Ana 2013; Santa Ana & Martino, 2009). Designed for dually diagnosed patients, a focus of the intervention is to examine the relationship between the substance use and the co-existing psychiatric disorder(s) and the importance of proactively treating both conditions.
  Arms: Arm 1 GMI
Behavioral: Arm 2 IHMD — Participants randomized to IHMD received a 27 day VA Care Coordination Home Telehealth (CCHT) program targeting acute recovery from alcohol and other drug disorders. IHMD consisted of daily assessment combined with dialogues consisting of motivational interviewing, cognitive behavioral therapy, and 12-step (mutual self-help) facilitation.
  Arms: Arm 2 IHMD
Behavioral: Arm 3 TCC — TCC consisted of a 4-session psychoeducational group (75 minutes per session). Material was delivered using a power point presentation on topics

SUMMARY:
Two approaches for providing evidence-based substance abuse treatment (EBT), group motivational interviewing (GMI) and the In-Home-Messaging-Device (IHMD), are interventions that have the characteristic ability for increasing accessibility to evidence-based treatment among patients with substance use problems and are proposed for investigation. GMI is based on motivational interviewing, an intervention that has shown consistent significant effects in promoting treatment retention and reduced substance use among individuals with substance use disorders, and is delivered in a group format. IHMD is a user-friendly computerized Tele-mental Health communication tool that allows interaction through the telephone line between a Veteran and the health care provider in an individual's home or residential placement. The current proposal aims to determine whether GMI and IHMD lead to a significantly greater increase in treatment engagement and reduction in alcohol use compared to a treatment control condition (TCC) among Veterans with a substance use problem and a co-existing psychiatric disorder.

DETAILED DESCRIPTION:
Dually diagnosed Veterans (N = 178) will be recruited from the Charleston, SC VAMC Outpatient Substance Abuse Treatment Center (SATC) and block randomized to TAU, GMI, or IHMD. Patients with alcohol dependence or abuse (including drug abuse) and a nonsubstance-related major Axis I disorder (e.g., bipolar disorder, depression, psychotic disorder) will be eligible for the study. Participants, who were referred to the study at time of triage or during the orientation phase of SATC, will be evaluated at baseline and approximately at a 1 and 3-month follow-up. Primary outcome measures will be alcohol use and treatment utilization as measured by number of days of alcohol use, number of binge alcohol drinking days, and quantity of alcohol consumed (in standard drinks, or SECs), and treatment attendance sessions based on objective CPRS patient medical records (i.e., number of all substance abuse outpatient, other mental health [e.g., PTSD, depression], and other substance abuse treatment sessions), and self-reported 12-step (number of self-help AA/NA) sessions, including days consulting with a 12-step or mutual self-help sponsor. Exploratory outcomes measures include number of illicit drug use days (e.g., cocaine, crack, marijuana, opiates, and sedatives).

Primary questions:

A. Does GMI lead to a significantly greater reduction in alcohol use and an increase in treatment engagement outcomes in the 3-month follow-up period compared to participants assigned to TCC?

Hypothesis: Participants who receive GMI will consume less alcohol and will be engaged in and attend more continuous treatment than participants in TCC in the 3-month follow-up period.

B. Does IHMD lead to a significantly greater reduction in alcohol use and an increase in treatment engagement outcomes in the 3-month follow-up period compared to participants assigned to TCC?

Hypothesis: Participants who receive IHMD will consume less alcohol and will be engaged in and attend more continuous treatment than participants in TCC in the 3-month follow-up period.

Exploratory question:

Compared to TCC, will GMI and IHMD lead to significantly fewer days of illicit drug use by 3-month follow-up?

Hypothesis: Compared to TCC, GMI and IHMD will result in a significant reduction in days of illicit drug use by 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide informed consent
* reading level at least at the 5th grade level
* ability to identify at least one collateral contact
* ability to be contacted by telephone at follow-up
* access to a working telephone line in the home or residential placement
* alcohol use or alcohol and drug use in the 28 days prior to hospitalization and current alcohol dependence (or abuse) or alcohol and drug abuse

Exclusion Criteria:

* auditory or visual impairment that would interfere with study procedures
* scheduled for discharge within 72 hours of initial screening
* diagnosis of dementia
* inability to speak or understand English
* unable to access a landline telephone for the IHMD treatment group

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-05-03 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. Santa Ana, PhD MA BA, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Price KL, Baker NL, McRae-Clark AL, Saladin ME, Desantis SM, Santa Ana EJ, Brady KT. A randomized, placebo-controlled laboratory study of the effects of D-cycloserine on craving in cocaine-dependent individuals. Psychopharmacology (Berl). 2013 Apr;226(4):739-46. doi: 10.1007/s00213-011-2592-x. Epub 2012 Jan 11. PMID 22234379
- [Result] Prisciandaro JJ, Myrick H, Henderson S, McRae-Clark AL, Santa Ana EJ, Saladin ME, Brady KT. Impact of DCS-facilitated cue exposure therapy on brain activation to cocaine cues in cocaine dependence. Drug Alcohol Depend. 2013 Sep 1;132(1-2):195-201. doi: 10.1016/j.drugalcdep.2013.02.009. Epub 2013 Mar 14. PMID 23497788
- [Result] Santa Ana EJ, Stallings DL, Rounsaville BJ, Martino S. Development of an in-home telehealth program for outpatient veterans with substance use disorders. Psychol Serv. 2013 Aug;10(3):304-314. doi: 10.1037/a0026511. Epub 2011 Dec 12. PMID 23937090

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 GMI: Participants in GMI first completed a baseline assessment, then returned 1 week later to attend four GMI sessions, each session lasting 75 minutes, administered on four consecutive days within the same week period. One and three months after the day of IRB consent, participants were provided 1 one-month and a 3-month follow-up, respectively.
- Arm 2 IHMD: Participants in IHMD first completed a baseline assessment, then received within a 1 week period their IHMD CCHT device to be used on a daily basis for 27 days in their home. One and three months after the day of IRB consent, participants were provided 1 one-month and a 3-month follow-up, respectively.
- Arm 3 TCC: Participants in TCC first completed a baseline assessment, then returned 1 week later to attend four TCC sessions, each session lasting 75 minutes, administered on four consecutive days within the same week period. One and three months after the day of IRB consent, participants were provided 1 one-month and a 3-month follow-up, respectively.
Period: Overall Study
Arm/Group | Arm 1 GMI | Arm 2 IHMD | Arm 3 TCC
Started | 59 | 62 | 59
Completed | 51 | 57 | 51
Not Completed | 8 | 5 | 8
Not completed — Lost to Follow-up | 2 | 3 | 2
Not completed — Withdrawal by Subject | 4 | 2 | 5
Not completed — In Jail | 1 | 0 | 1
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 GMI: Group Motivational Interviewing
- Arm 2 IHMD: In-Home-Messaging Device
- Arm 3 TCC: Treatment Control condition
- Total: Total of all reporting groups
Arm/Group | Arm 1 GMI | Arm 2 IHMD | Arm 3 TCC | Total
Number analyzed (Participants) | 59 | 62 | 59 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (8.8) | 52.3 (10.3) | 51.1 (10.6) | 52.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 14
  Male | 54 | 58 | 54 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 32 | 36 | 36 | 104
  White | 27 | 25 | 22 | 74
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 59 | 62 | 59 | 180

OUTCOME MEASURES:

1. Primary Outcome: Number of Alcohol Drinking Days in the Previous 30 (One Month Follow up) and 60 (Three Month Follow up) Days
Description: Number of alcohol drinking days is the number of days that that participant self-reported having at least 1 standard alcohol beverage during the specified follow up period on the Time Line Follow Back (Sobell & Sobell, 1992).
Time Frame: One month follow-up and three month follow up in the previous 30 (one month follow up) and 60 (three month follow up) days
Population: Intent to treat population (at least one GMI session attended)
Measure: Mean (Standard Deviation); unit: Days Using Alcohol
Groups:
- Arm 2 IHMD: In Home Messaging Device
Arm/Group | Arm 1 GMI | Arm 2 IHMD | Arm 3 TCC
Number analyzed (Participants) | 59 | 62 | 59
Days Using Alcohol
  One month follow up | 5.1 (7.6) | 6.5 (9.5) | 6.7 (10.3)
  Three month follow up | 8.8 (13.3) | 10.9 (16.3) | 9.9 (18.8)
Statistical Analysis 1: Comparison: Arm 1 GMI vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — Zero-inflated Poisson model with random intercept to account for correlation between repeated measurements of the responses within subjects was conducted; p < 0.01, Zero inflated Poisson model
Statistical Analysis 2: Comparison: Arm 2 IHMD vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — Zero-hurdle Poisson model with random intercept to account for correlation between repeated measurements of the responses within subjects was conducted; p = 0.02, zero-hurdle Poisson model

2. Primary Outcome: Number of Alcohol Binge Drinking Days in the Previous 30 (One Month Follow up) and 60 (Three Month Follow up) Days
Description: Number of alcohol binge drinking days is the number of days that that participant self-reported having at least 4 standard alcohol beverages on one occasion (for women) and at least 5 standard alcohol beverages on one occasion (for men) during the specified follow up period on the Time Line Follow Back (Sobell & Sobell, 1992).
Time Frame: One and three-months post intervention in the previous 30 (one month follow up) and 60 (three month follow up) days
Population: Intent to treat population (at least one GMI session attended)
Measure: Mean (Standard Deviation); unit: Days of binge drinking
Groups:
- Arm 2 (IHMD): In-Home-Messaging-Device
Arm/Group | Arm 1 GMI | Arm 2 (IHMD) | Arm 3 TCC
Number analyzed (Participants) | 59 | 62 | 59
Days of binge drinking
  One month follow up | 3.1 (6.5) | 2.7 (6.5) | 6.1 (10.5)
  Three month follow up | 5.1 (10.8) | 4.0 (10.5) | 7.9 (17.7)
Statistical Analysis 1: Comparison: Arm 1 GMI vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — A Zero-inflated Poisson model with random intercept to account for correlation between repeated measurements of the responses within subjects was conducted; p < 0.01, Zero inflated Poisson model
Statistical Analysis 2: Comparison: Arm 2 (IHMD) vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = .0002, Zero-hurdle Poisson model

3. Primary Outcome: Standard Number of Alcohol Drinks in the Previous 30 (One Month Follow up) and 60 (Three Month Follow up) Days
Description: Standard drinks, or SECs, is the number of drinks that the participant self-reported consuming (as measured by 0.5 oz ethanol alcohol per beverage) during the specified follow up period on the Time Line Follow Back (Sobell & Sobell, 1992).
Time Frame: One and three-months post intervention in the Previous 30 (One Month Follow up) and 60 (Three Month Follow up) Days
Population: Intent to treat population (at least one GMI session attended)
Measure: Mean (Standard Deviation); unit: Standard alcohol drinks
Arm/Group | Arm 1 GMI | Arm 2 (IHMD) | Arm 3 TCC
Number analyzed (Participants) | 59 | 62 | 59
Standard alcohol drinks
  One month follow up | 45.1 (98.1) | 45.8 (100.7) | 70.0 (131.1)
  Three month follow up | 66.5 (156.6) | 64.6 (129.7) | 112.3 (251.9)
Statistical Analysis 1: Comparison: Arm 1 GMI vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — To examine differences between GMI and TCC on SECs, a two-component Weibull mixture model for effectively dealing with zero-heavy continuous data was conducted; p = 0.04, Weibull mixture model
Statistical Analysis 2: Comparison: Arm 2 (IHMD) vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — A generalized linear mixed model with correlated errors to account for correlation between repeated measurements of the response within subjects was conducted; p = 0.47, Mixed Models Analysis

4. Primary Outcome: Treatment Utilization in the Previous 30 (One Month Follow up) and 60 (Three Month Follow up) Days
Description: Treatment utilization is the number of treatment attendance sessions based on objective CPRS medical records, including number of all VA substance abuse outpatient, other mental health (e.g., PTSD, depression), and other substance abuse treatment sessions.
Time Frame: One and three-months post intervention in the Previous 30 (One Month Follow up) and 60 (Three Month Follow up) Days
Population: Intent to treat population (at least one GMI session attended)
Measure: Mean (Standard Deviation); unit: Number of treatment sessions
Arm/Group | Arm 1 GMI | Arm 2 (IHMD) | Arm 3 TCC
Number analyzed (Participants) | 59 | 62 | 59
Number of treatment sessions
  One month follow up | 8.7 (8.7) | 7.0 (9.6) | 8.8 (9.0)
  Three month follow up | 11.3 (13.2) | 6.4 (9.8) | 8.3 (11.1)
Statistical Analysis 1: Comparison: Arm 1 GMI vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — Zero inflated Poisson model with random intercept to account for correlation between repeated measurement of the responses within subjects was conducted; p < 0.01, Zero inflated Poisson model
Statistical Analysis 2: Comparison: Arm 2 (IHMD) vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p < .0001, Zero-hurdle Poisson model

5. Primary Outcome: Treatment Attendance at 12-step or Mutual Self-help Sessions in the Previous 30 (One Month Follow up) and 60 (Three Month Follow up) Days
Description: Number of self-reported 12-step (number of self-help alcoholics anonymous or narcotics anonymous [AA/NA]) sessions, including days of consulting with a 12-step sponsor for help with a substance use problem based on the Time Line Follow-Back (Sobell & Sobell, 1992).
Time Frame: One and three-months post intervention in the Previous 30 (One Month Follow up) and 60 (Three Month Follow up) Days
Population: Intent to treat population (at least one GMI session attended)
Measure: Mean (Standard Deviation); unit: Number of 12-step sessions attended
Arm/Group | Arm 1 GMI | Arm 2 (IHMD) | Arm 3 TCC
Number analyzed (Participants) | 59 | 62 | 59
Number of 12-step sessions attended
  One month follow up | 8.0 (12.0) | 5.1 (8.8) | 7.1 (29.6)
  Three month follow up | 16.2 (22.4) | 10.6 (16.6) | 16.2 (22.4)
Statistical Analysis 1: Comparison: Arm 1 GMI vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < .0001, Zero inflated Poisson model
Statistical Analysis 2: Comparison: Arm 2 (IHMD) vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.02, Zero-hurdle Poisson model

6. Secondary Outcome: Number of Illicit Drug Use Days in the Previous 30 (One Month Follow up) and 60 (Three Month Follow up) Days
Description: Number of illicit drug use days is the number of days that that participant self-reported having used illicit drug (e.g., cocaine, crack, marijuana, opiates, sedatives, hallucinogens) during the specified follow up period on the Time Line Follow Back (Sobell & Sobell, 1992).
Time Frame: One and three-months post intervention in the Previous 30 (One Month Follow up) and 60 (Three Month Follow up) Days
Population: Intent to treat population (at least one GMI session attended)
Measure: Mean (Standard Deviation); unit: Days of drug use
Arm/Group | Arm 1 GMI | Arm 2 (IHMD) | Arm 3 TCC
Number analyzed (Participants) | 59 | 62 | 59
Days of drug use
  One month follow up | 0.74 (1.6) | 0.62 (2.3) | 0.7 (1.6)
  Three month follow up | 0.9 (2.0) | 0.51 (1.6) | 0.7 (2.0)
Statistical Analysis 1: Comparison: Arm 1 GMI vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.17, Zero inflated Poisson model
Statistical Analysis 2: Comparison: Arm 2 (IHMD) vs Arm 3 TCC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; p = 0.67, Zero-hurdle Poisson model

ADVERSE EVENTS:
Arm/Group | Arm 1 GMI | Arm 2 IHMD | Arm 3 TCC
Serious Adverse Events (participants affected / at risk) | 2/59 | 0/62 | 0/59
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 GMI (N=59) | Arm 2 IHMD (N=62) | Arm 3 TCC (N=59)
Suicidal Ideation (Psychiatric disorders) | 1 (59) | 0 (0) | 0 (0) — A participant indicated positively that he was experiencing suicidal ideation. Participant was evaluated by a VA psychiatrist who determined that the patient should be hospitalized for stabilization. This was reported to the IRB.
Death due to throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (59) | 0 (0) | 0 (0) — Participant had throat cancer and died during follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No